CLINICAL TRIAL: NCT01423227
Title: Benefits and Costs of Home-based Pulmonary Rehabilitation in Chronic Obstructive Pulmonary Disease
Acronym: HomeBase
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: La Trobe University (Other)
Collaborators: The Alfred (Other); Austin Health (Other Government); Monash University (Other)
Responsible Party: Principal Investigator, Anne Holland, Associate Professor, La Trobe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HomeBase
Record Dates: First submitted 2011-08-11; First posted 2011-08-25 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; exercise; rehabilitation; dyspnea; quality of life; economic evaluation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity; Dyspnea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Home-based pulmonary rehabilitation (Experimental): Home visit plus 8 weeks of once-weekly telephone calls
  Interventions: Behavioral: Home-based pulmonary rehabilitation
- Hospital-based pulmonary rehabilitation (Active Comparator): Standard twice-weekly 8-week outpatient pulmonary rehabilitation program
  Interventions: Behavioral: Hospital-based pulmonary rehabilitation

INTERVENTIONS:
Behavioral: Home-based pulmonary rehabilitation — One home visit plus weekly telephone calls for 8 weeks
  Arms: Home-based pulmonary rehabilitation
Behavioral: Hospital-based pulmonary rehabilitation — Standard twice-weekly 8-week outpatient pulmonary rehabilitation program
  Arms: Hospital-based pulmonary rehabilitation

SUMMARY:
Pulmonary rehabilitation is an effective treatment for people with chronic obstructive pulmonary disease (COPD) which improves symptoms, reduces hospitalisation and lowers healthcare costs. However less than 1% of Australians with COPD receive pulmonary rehabilitation each year, due to poor access to programs and high levels of disability. This randomised controlled trial will examine the benefits and costs of a novel, entirely home-based pulmonary rehabilitation program for COPD. We hypothesise that home-based pulmonary rehabilitation can deliver equivalent clinical outcomes at lower cost than the centre-based program.

We will randomly allocate 144 people with COPD to undertake either standard pulmonary rehabilitation in a hospital setting, or a low-cost home-based program. Those who undertake pulmonary rehabilitation in the hospital setting will attend the hospital twice each week for eight weeks for supervised exercise training and education. People in the home pulmonary rehabilitation group will receive one home visit and weekly telephone calls for eight weeks, for supervision and mentoring of exercise and provision of education. We will compare the number of people who complete the program in each setting. We will also test whether the groups have similar results for the standard pulmonary rehabilitation outcomes of breathlessness, quality of life and exercise capacity, at the end of the program and 12 months later. We will compare health care costs and personal costs between groups after 12 months.

If home-based pulmonary rehabilitation can improve uptake of this important treatment, deliver good clinical outcomes and reduce costs this will have significant and long-lasting benefits for patients, the community and the health system

ELIGIBILITY:
Inclusion Criteria:

* current or former smokers of at least 10 packet years
* aged 40 years or over
* diagnosis of COPD confirmed on spirometry.

Exclusion Criteria:

* previous diagnosis of asthma
* have attended a pulmonary rehabilitation program in the last two years
* exacerbation of COPD within the last four weeks
* have comorbidities which prevent participation in an exercise training program

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2011-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in 6-minute walk test | Baseline, 8 weeks and 12 months
  Testing equivalence between groups

SECONDARY OUTCOMES:
Change in Chronic Respiratory Disease Questionnaire | Baseline, 8 weeks and 12 months
Change in Modified Medical Research Council Scale | Baseline, 8 weeks and 12 months
Cost-effectiveness | 12 months
SF-36 v2 | Baseline, 8 weeks and 12 months
  Contributes to cost effectiveness analysis
Program completion rate | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anne E Holland, PhD, Principal Investigator — La Trobe University, Alfred Health, Institute for Breathing and Sleep; Christine F McDonald, PhD, Principal Investigator — Austin Health, Institute for Breathing and Sleep; Ajay Mahal, PhD, Principal Investigator — Monash University
Locations (2):
- Australia (2):
  - Austin Health, Heidelberg, Victoria
  - Alfred Health, Melbourne, Victoria

REFERENCES:
- [Derived] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633
- [Derived] Grimwood CL, Holland AE, McDonald CF, Mahal A, Hill CJ, Lee AL, Cox NS, Moore R, Nicolson C, O'Halloran P, Lahham A, Gillies R, Burge AT. Comparison of self-report and administrative data sources to capture health care resource use in people with chronic obstructive pulmonary disease following pulmonary rehabilitation. BMC Health Serv Res. 2020 Nov 23;20(1):1061. doi: 10.1186/s12913-020-05920-0. PMID 33228654
- [Derived] Burge AT, Holland AE, McDonald CF, Abramson MJ, Hill CJ, Lee AL, Cox NS, Moore R, Nicolson C, O'Halloran P, Lahham A, Gillies R, Mahal A. Home-based pulmonary rehabilitation for COPD using minimal resources: An economic analysis. Respirology. 2020 Feb;25(2):183-190. doi: 10.1111/resp.13667. Epub 2019 Aug 16. PMID 31418515
- [Derived] Hoaas H, Zanaboni P, Hjalmarsen A, Morseth B, Dinesen B, Burge AT, Cox NS, Holland AE. Seasonal variations in objectively assessed physical activity among people with COPD in two Nordic countries and Australia: a cross-sectional study. Int J Chron Obstruct Pulmon Dis. 2019 Jun 5;14:1219-1228. doi: 10.2147/COPD.S194622. eCollection 2019. PMID 31239657
- [Derived] Lahham A, McDonald CF, Mahal A, Lee AL, Hill CJ, Burge AT, Cox NS, Moore R, Nicolson C, O'Halloran P, Gillies R, Holland AE. Participation in Physical Activity During Center and Home-Based Pulmonary Rehabilitation for People With COPD: A SECONDARY ANALYSIS OF A RANDOMIZED CONTROLLED TRIAL. J Cardiopulm Rehabil Prev. 2019 Mar;39(2):E1-E4. doi: 10.1097/HCR.0000000000000373. PMID 30688793
- [Derived] Liacos A, McDonald CF, Mahal A, Hill CJ, Lee AL, Burge AT, Moore R, Nicolson C, O'Halloran P, Cox NS, Lahham A, Gillies R, Holland AE. The Pulmonary Rehabilitation Adapted Index of Self-Efficacy (PRAISE) tool predicts reduction in sedentary time following pulmonary rehabilitation in people with chronic obstructive pulmonary disease (COPD). Physiotherapy. 2019 Mar;105(1):90-97. doi: 10.1016/j.physio.2018.07.009. Epub 2018 Aug 3. PMID 30316548
- [Derived] Holland AE, Mahal A, Hill CJ, Lee AL, Burge AT, Cox NS, Moore R, Nicolson C, O'Halloran P, Lahham A, Gillies R, McDonald CF. Home-based rehabilitation for COPD using minimal resources: a randomised, controlled equivalence trial. Thorax. 2017 Jan;72(1):57-65. doi: 10.1136/thoraxjnl-2016-208514. Epub 2016 Sep 26. PMID 27672116
- [Derived] Holland AE, Mahal A, Hill CJ, Lee AL, Burge AT, Moore R, Nicolson C, O'Halloran P, Cox NS, Lahham A, Ndongo R, Bell E, McDonald CF. Benefits and costs of home-based pulmonary rehabilitation in chronic obstructive pulmonary disease - a multi-centre randomised controlled equivalence trial. BMC Pulm Med. 2013 Sep 8;13:57. doi: 10.1186/1471-2466-13-57. PMID 24011178